CLINICAL TRIAL: NCT06920134
Title: Study on Preliminary Safety and Efficacy of the ARC-IM Therapy to Support Hemodynamic Management in People With Typical and Atypical Parkinson's Disease
Brief Title: Epidural Electrical Stimulation to Support Hemodynamic Management in Individuals With Parkinson's Disease
Acronym: PD-HemON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Principal Investigator, Jocelyne Bloch, Professor, Centre Hospitalier Universitaire Vaudois
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD-HemON; HT94252410901 (Other Grant/Funding Number: Department of Defense, USAMRAA); CDMRP-PD230100 (Other Grant/Funding Number: CDMRP-Proposal Log Number)
Record Dates: First submitted 2025-03-24; First posted 2025-04-09 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-07

CONDITIONS: Hypotension Symptomatic; Parkinson's Disease; Orthostatic Hypotension, Dysautonomic; Multiple System Atrophy (MSA) With Orthostatic Hypotension; Multiple System Atrophy - Parkinsonian Subtype (MSA-P)
Keywords: orthostatic hypotension; parkinson's disease; autonomic failure; hypotension
MeSH Terms: conditions — Parkinson Disease; Shy-Drager Syndrome; Multiple system atrophy (MSA) with orthostatic hypotension; Hypotension, Orthostatic; Pure Autonomic Failure; Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): All participants will be provided with the ARC-IM Investigational System (implantable and non-implan
  Interventions: Device: ARC-IM Investigational System

INTERVENTIONS:
Device: ARC-IM Investigational System — Implantation of a stimulation lead on the low thoracic level of the spinal cord and implantation of a neurostimulator in the abdominal region.

SUMMARY:
The PD-HemON study aims to evaluate the safety and preliminary efficacy of ARC-IM Therapy (Epidural Electrical Stimulation) to support hemodynamic management in people with typical and atypical Parkinson's Disease, who suffer from orthostatic hypotension.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years old
2. Typical or Atypical PD (including but not limited to Multiple System Atrophy, Pure Autonomic Failure, Progressive Supranuclear Palsy)
3. Confirmed orthostatic hypotension with a test for verticalization
4. Confirmed symptomatic orthostatic hypotension that makes daily activities particularly challenging as determined by the study clinicians
5. Must provide and sign the Informed Consent before any study-related procedures
6. Stable medical, physical, and psychological conditions given participant indication as considered by Investigators;
7. Able to understand and interact with the study team in French or English
8. Agrees to comply in good faith with all conditions of the study and to attend all scheduled appointments

Exclusion Criteria:

1. Diseases and conditions that would increase the morbidity and mortality of the implantation surgery
2. The inability to withhold antiplatelet/anticoagulation agents perioperatively
3. History of myocardial infarction or cerebrovascular events within the past 6 months
4. Unstable or significant medical condition that is likely to interfere with study procedures or likely to confound study endpoint evaluations as determined by the Investigator
5. History or presence of major psychiatric disorders or major neurocognitive disorders as considered by the Investigators in accordance with the treating physician and treating neurologist
6. Major changes in PD treatment planned until the end of the main study phase (such as DBS or dopamine-pump implantation)
7. Inability to follow study procedures.
8. Spinal anatomical abnormalities precluding surgery
9. Presence of any indications requiring frequent MRIs.
10. Current pregnancy or current breastfeeding
11. Lack of effective or acceptable contraception for women of childbearing capacity
12. Intention to become pregnant during the study
13. Unable or unwilling to effectively use the study system or related devices by the participant or caretaker, as determined by the investigator
14. Participation in another interventional study that might confound study endpoint evaluations
15. Enrolment of the investigator, his/her family members, employees, and other dependent persons

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2031-05-01 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of (serious) adverse device effects of the ARC-IM Therapy from baseline up to the end of the study. | Throughout the study (up to 5 years)
  Evaluate the safety of ARC-IM Therapy in supporting hemodynamic management in participants with atypical or typical Parkinson's Disease and orthostatic hypotension

SECONDARY OUTCOMES:
10-minute, orthostatic head-up tilt test with and without the ARC-IM Therapy at 1 month after intervention | At the end of, 6 months after and 1 year after configuration of the therapy,
  Preliminary and long-term efficacy of the ARC-IM Therapy to reduce orthostatic hypotension.
  Measurement tool: Drop in blood pressure over time (mmHg and sec, mmHg/sec)
Severity of symptoms measured by The Orthostatic Hypotension Questionnaire. | At the end of, 6 months after and 1 year after configuration of the therapy
  This outcome measures the preliminary long-term efficacy of the ARC-IM Therapy to support hemodynamic instability. The Orthostatic Hypotension Questionnaire (OHQ) has 10 hypotension symptom-related items rated on a 11 point scale (0 - 10).
  Measurement tool: 0 indicates no symptoms and 10 indicates worst possible severity/outcome. A higher total score indicates worse symptomatology.
Time Up and Go Test (TUG) | At the end of, 6 months after and 1 year after configuration of the therapy
  Preliminary efficacy of the ARC-IM Therapy to improve physical activity. The Time Up and Go will measure time from sit to stand and gait quality. Measurement tool: time (sec)
2 Minute Walk Test | At the end of, 6 months after and 1 year after configuration of the therapy
  Preliminary efficacy of the ARC-IM Therapy to improve physical activity. The 2 Minute Walk Test (2MWT) will measure gait endurance and distance walked over 2 minutes.
  Measurement tool: distance (meters)
Berg Balance Test | At the end of, 6 months after and 1 year after configuration of the therapy
  The Berg Balance Test measures the ability to balance safely with 14 specific tasks performed while standing, sitting, or making simple movements. The test scoring ranges from 0 to 56.
  Measurement tool: lower score indicates greater risk of losing your balance.
Quebec User Evaluation of Satisfaction with technology (QUEST 2.0) | At 6 months and 1 year after configuration of the therapy
  To measure the usability of the ARC-IM Main Controller, Clinician Programmer, and Personal Programmer for clinicians and participants.
  The Quebec User Evaluation of Satisfaction with technology (QUEST 2.0) is a 12-item instrument that evaluates satisfaction with the therapy across form factor, safety, durability, simplicity of use, comfort, service of device and improvements. The evaluation will be performed by a moderator with the participant.
  Measurement tool: Total score from 12 to 60. Low score means a better outcome.
System Usability Scale (SUS) | At 6 months and 1 year after configuration of the therapy
  Assess the usability of the ARC-IM Main Controller, Clinician Programmer, and Personal Programmer for clinicians and participants.
  The System Usability Scale (SUS) is a 10-item scale that evaluates the usability and satisfaction of the technology.
  Measurement tool: Total score from 0 to 100. Higher score indicates better outcome.
Additional user feedback of ARC-IM System | At 6 months and 1 year after configuration of the therapy
  To assess the usability of the ARC-IM Main Controller, Clinician Programmer, and Personal Programmer for clinicians and participants.
  The Additional user feedback of ARC-IM System is a custom-made user feedback questionnaire to evaluate the overall satisfaction of specific aspects of the therapy including battery life, device communication etc.
  Measurement tool: Total score where applicable (higher score indicates better outcome) and feedback from participants

OTHER OUTCOMES:
Doppler ultrasound to measure cerebral blood perfusion with and without the ARC-IM Therapy | 1 month, 6 months and 12 months post-therapy configuration
Supine hypertension will be evaluated during orthostatic tilt tests without the ARC-IM Therapy | 1 month, 6 months and 12 months post-therapy configuration
  Measurement tool: blood pressure (mmHg) during supine position of orthostatic tilt test
MDS-sponsored Unified Parkinson's Disease Rating Scale Part IB & II | 1 month, 6 months and 12 months post-therapy configuration
  Participants' quality of life will be assessed with MDS-sponsored Unified Parkinson's Disease Rating Scale Part IB & II to measure sleep, mental health, and fatigue (MDS-UPDRS-IB & II) over 20 items.
  Measurement tool: Total score (0 - 4 rating per question), 0 represents no impairment and 4 represents severe impairment. Higher total score indicates worse symptoms.
King's Parkinson's Disease Pain Scale | 1 month, 6 months and 12 months post-therapy configuration
  Participants' quality of life will be assessed with the 7-item King's Parkinson's Disease Pain Scale to characterize severity and types of pain associated with Parkinson's Disease.
  Measurement tool: Total score from 0 to 168. Lower score indicates a better outcome.
Parkinson's Disease Questionnaire-39 (PDQ-39) | 1 month, 6 months and 12 months post-therapy configuration
  Participants' quality of life will be measured by the 39 item Parkinson's Disease Questionnaire-39 (PDQ-39) to evaluate perceived health in terms of physical, mental and social functions.
  Measurement tool: Total score from 0-100, higher scores reflect lower quality of life
Scales for Outcomes in Parkinson's disease - Autonomic Dysfunction | 1 month, 6 months and 12 months post-therapy configuration
  Scales for Outcomes in Parkinson's disease - Autonomic Dysfunction (SCOPA-AUT) is a 25-item, self-completed questionnaire to evaluate autonomic symptoms in people with typical and atypical Parkinson's Disease.
  Measurement tool: Total score from 0-69 where a higher score indicates increased frequency of autonomic dysfunction symptoms
MDS sponsored Unified Parkinson's Disease Rating Scale Part III | Baseline (before surgery), and 1 month, 6 months and 12 months post-therapy configuration
  Participants' quality of life will be assessed with the MDS-sponsored Unified Parkinson's Disease Rating Scale Part III (19 items) to evaluate motor function.
  Measurement tool: Total score from 0 to 132. Low score means a better outcome.
24 hour ambulatory measurements | Baseline (before surgery), and 1 month, 6 months and 12 months post-therapy configuration
  Participant's quality of life will be evaluated with 24 hour blood pressure measurements with and without the therapy.
  Measurement tool: blood pressure (mmHg)
Closed-loop stimulation on management of hemodynamics will be measured with the change in blood pressure during 10 minute, head up tilt tests. | Post-operative configuration phases, through year 1 of the study
  Closed-loop stimulation will receive feedback from a blood pressure sensor to automatically adjust stimulation intensity. We will evaluate the effects of this stimulation on management of hemodynamics during configuration sessions with pre-configured stimulations, with closed-loop stimulation and without stimulation. The feasibility and effectiveness will be measured by the drop in blood pressure (mmHg) during 10 minute, orthostatic, head-up tilt tests.
Time Up and Go Test across different therapeutic conditions | Post-operative configuration phases, through year 1 of the study
  The complementarity of the ARC-IM Therapy with standard therapies (e.g LDopa) will be assessed over the trajectory of therapy intake with and without stimulation during configuration phases with the Time Up and Go will measure time from sit to stand and gait quality.
  Measurement tool: time (sec)
2 Minute Walk Test across different therapeutic conditions | Post-operative configuration phases, through year 1 of the study
  The complementarity of the ARC-IM Therapy with standard therapies (e.g LDopa) will be assessed over the trajectory of therapy intake with and without stimulation during configuration phases with the The 2 Minute Walk Test (2MWT) will measure gait endurance and distance walked over 2 minutes.
  Measurement tool: distance (meters)
Berg Balance Test across different therapeutic conditions | Post-operative configuration phases, through year 1 of the study
  The complementarity of the ARC-IM Therapy with standard therapies (e.g LDopa) will be assessed over the trajectory of therapy intake with and without stimulation during configuration phases with the Berg Balance Test measures the ability to balance safely with 14 specific tasks performed while standing, sitting, or making simple movements.
  Measurement tool: Total score from 0-56, lower score indicates greater risk of losing your balance.

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyne Bloch, MD, Principal Investigator — CHUV
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland